CLINICAL TRIAL: NCT01714557
Title: Piperacillin/Tazobactam for Prophylaxis in Patients of Neutropenia After Hematopoietic Stem Cell Transplantation - A Pilot Study
Brief Title: Prophylactic Piperacillin/Tazobactam in Hematopoietic Stem Cell Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Wenrong Huang, Associate director, Hematology, Chinese PLA General hospital, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TZP-HEM-20120608
Record Dates: First submitted 2012-07-04; First posted 2012-10-26 (Estimated); Last update posted 2012-10-26 (Estimated); Status verified 2012-10

CONDITIONS: Neutropenia; Hematopoietic Stem Cell Transplantation
MeSH Terms: conditions — Neutropenia | interventions — Piperacillin; Piperacillin, Tazobactam Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- No prophylaxis (No Intervention)
- piperacillin (Active Comparator)
  Interventions: Drug: Piperacillin
- piperacillin/tazobactam (Experimental)
  Interventions: Drug: Piperacillin-tazobactam combination product

INTERVENTIONS:
Drug: Piperacillin — 4.0g q8h 3-5 days
  Arms: piperacillin
Drug: Piperacillin-tazobactam combination product — 4.5g q8h 3-5 days
  Other Names: Tazocin
  Arms: piperacillin/tazobactam

SUMMARY:
Neutropenia is very common in patients received hematopoietic stem cell transplantation, with median duration of about 14 days. Almost all neutropenia will suffer from febrile without prophylactic antibiotics. IDSA recommended fluoroquinolones as prophylaxis in neutropenia patients of high risks, while in China, major pathogens possess high resistance to fluoroquinolones. It is not clear whether prophylaxis is of benefit, nor the appropriate prophylaxis regimen.

The current study will evaluate the three different regimen:

1. No prophylaxic antibiotic
2. Piperacillin as prophylaxis for neutropenia patients. Piperacillin has anti-pseudomonas activity.
3. Piperacillin/tazobactam as prophylaxis for neutropenia patients. Piperacillin/tazobactam has highest susceptibility rate among common anti-pseudomonas antibiotics.

DETAILED DESCRIPTION:
1. Swab culture (skin, pharyngeal, nasal, anus) when administered into laminar flow room after transplantation.
2. Randomize the neutropenia patients into 3 groups.
3. Receive 3 regimen.
4. Full record of clinical data, including background diseases, previous antibiotics within 90 days, febrile or not at the TOC.
5. For patients developed febrile, imipenem will be prescribed, even if the patient received no prophylaxis. At the same time, the follow-up ended.

ELIGIBILITY:
Inclusion Criteria:

* Age 13-65 years
* Received Autologous or Allogeneic hematopoietic stem cell transplantation.
* ECOG score 0-1.
* ICF is available.

Exclusion Criteria:

* Allergic to any therapy drug.
* Documented infection before neutropenia.
* Renal dysfunction.
* Suffering from central nervous system or mental disease.

Ages: 13 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2012-09; Primary Completion 2014-09 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
febrile rate | 3 weeks after beginning of prophylaxis
  In both group, how many patients developed febrile.

SECONDARY OUTCOMES:
Microbiologic efficacy in febrile patients | 3 weeks after beginning of prophylaxis
  The success rate and failure rate will be calculated.
  1. The microbiologic culture is positive at 3 weeks of prophylaxis, showing pathogen sensitive to Piperacillin/tazobactam, the case will be evaluated as breakthrough infection, that means microbiologic failure.
  2. The microbiologic culture is negative at 3 weeks of prophylaxis,, or positive fungus or non-typical organisms, the case will be evaluated as microbiologic success.
Recovery rate from neutropenia | 3 weeks after beginning of prophylaxis
  How many patients reached the ANC > 0.5×109/L more than 3 days.
AE | 3 weeks after beginning of prophylaxis
  How many patients developed unexpected medical events.
Cost of drug and hospital-stay | 3 weeks after beginning of prophylaxis

CONTACTS AND LOCATIONS:
Overall Officials: wenrong huang, Doctor, Principal Investigator — Employee
Locations (1):
- Chinese PLA general hospital, Beijing, Beijing Municipality, China